CLINICAL TRIAL: NCT02910934
Title: Cost-effectiveness Evaluation of Vector Control Strategies in Mozambique
Acronym: COST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Abt Associates (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Mozambique (Other Government); Centro de Investigacao em Saude de Manhica (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 946238-1 (EOM)
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Malaria
Keywords: Indoor Residual Spray; IRS; Insecticide Treated Net; LLIN; ITN; Long lasting insecticidal net
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IRS (Experimental): This arm is comprised of village clusters that have received indoor residual spray with Actellic CS.
  Interventions: Other: Actellic CS
- non-IRS (No Intervention): This arm is comprised of village clusters that will not receive indoor residual spray

INTERVENTIONS:
Other: Actellic CS — Indoor residual spray with Actellic CS
  Arms: IRS

SUMMARY:
This study aims to provide National Malaria Control Programs (NMCP), international donors and other key stakeholders with clear evidence on the impact and cost-effectiveness of using indoor residual spraying (IRS) with a non-pyrethroid insecticide in a high malaria transmission area that has universal long-lasting insecticidal net (LLIN) coverage. This is an interventional study with IRS serving as the research intervention.

The district of Mopeia, in the province of Zambezia, Mozambique will be the study site. This is a high transmission area with a malaria parasite prevalence of 54% in children. The Ministry of Health distributed LLINs in Mopeia in 2014-2015.

The NMCP through funding from President's Malaria Initiative Africa Indoor Residual Spraying Project (PMI-AIRS) was able to cover half a district with indoor residual spraying. A simplified census took place in mid-2016 to determine the number of children five years of age and under in the district and enumerate and map the households to assist in implementation.

From the 115 villages/bairros existent in Mopeia, 86 clusters were randomized in a government randomization ceremony to either receive IRS with Actellic or maintain no IRS. The IRS was implemented through a partnership between the NMCP and PMI-AIRS according to standard operational and consent procedures. From each cluster, a cohort of 18 children five years of age and under will be followed monthly to assess malaria incidence at the community level in both IRS and non-IRS villages. There will be 774 children in the IRS villages and 774 children in the no-IRS villages (total cohort will be 1548). Additionally, the routine health centre reporting system will be strengthened to assess malaria incidence in children five years of age and under by passive case detection. Three cross sectional studies in April 2017, April 2018, and April 2019 will assess changes in net use, health seeking behaviour and malaria prevalence at the community level.

Entomological data will be collected from both IRS and non-IRS areas to assess the vector dynamics and insecticide resistance pattern of the local vector populations from sprayed and unsprayed areas. Data on the costs of the implementation as well as health-related expenditures at health system and household levels will be collected prospectively throughout the study. These costs will be determined using both health system and societal perspectives.

The incidence rate in IRS and no-IRS areas will be combined with the micro-costing data to calculate the cost per case averted at community and health facility level.

These findings will be disseminated to the NMCP and international donors and stakeholders to complement the World Health Organization (WHO) guidance on combining indoor residual spraying and long-lasting insecticidal nets.

DETAILED DESCRIPTION:
Mopeia is a district in the Zambezia Province. Mopeia borders the district of Morrumbala to the North, the district of Chinde and the province of Sofala to the South, the districts of Nicoadala and Inhassunge in the East and the Provinces of Sofala and Tete in the West. It has an area of 7671 km2. The projected population for 2016 is 162.188 individuals with 31.927 (19.7%) under five years of age (National Institute of Statistics, Mozambique). There are three administrative posts, eleven localities and 224 villages (Bairros) and approximately 34.603 households. There are 12 health facilities (PMI-AIRS Mozambique, unpublished data). There is little socio-economic data available from Mopeia.

The malaria burden is high in Zambezia with a parasite prevalence of 54% in under-fives [19]. The parasite prevalence in children 1-15 years of age in Mopeia is 47.8% (38.7%-57.1%) [20]. The mean rapid diagnostic test (RDT) positivity rate during a recent enhanced surveillance exercise at health facilities was 62.8% (range 50-72%) [21]. The same data suggest high incidence at health facilities, showing 470 cases per 1000 children during the same period (June-Nov 2014). Mopeia recently received 175.297 LLINs in 2013 and IRS with pyrethroids in 2014 [22]. Residents of Mopeia will receive new LLINs in early 2017.

Data from February 2015 in the neighbouring districts of Mocuba and Morrumbala show Pyrethroid resistance in the local Anopheles gambiae s.l. population [23]. Further north, in the district of Milange, tested Anopheles gambiae s.l. remain susceptible to pyrethroids [23]. See table 2 below for further details. Mopeia has been selected to receive IRS because of its high malaria transmission intensity, the presence of LLINs in the district, and the aforementioned regional indications of reduced pyrethroid susceptibility in the target vector population, and the existence of IRS infrastructure and capacity from previous campaigns.

The villages selected for spraying will receive IRS with Actellic according to standard operating and consent procedures [24] in addition to existing LLINs. Non IRS areas will have existing LLINs, but will not receive IRS. In late 2017 (year two), IRS will be repeated using the same village selection and insecticide. Additionally in 2017, the whole district will be subject to universal LLIN distribution.

Individuals enrolled in the cohort were recruited independent of their household acceptance or refusal of spray. IRS status will be confirmed with questionnaires during the monthly active cohort visits and during the cross-sectional surveys, including questions about wall replastering/painting and net usage (SSPs COST 001, 002 and 003). Additional information will be obtained through cone bioassays.

The standard of malaria care at community and health center will remain unchanged throughout the study and stock levels of malaria commodities will be ensured.

This study of IRS implementation in Mozambique will provide detailed information of the impact and cost-effectiveness of adding IRS with an extended release formulation of the organophosphate insecticide pirimiphos-methyl (Actellic®300CS) in a high transmission area with high LLIN coverage. This information will be disseminated to the NMCP as well as to local and international stakeholders and decision makers to inform policy recommendations and choices regarding the combination of vector control strategies.

A simplified census was conducted in June-July 2016 to obtain the total number of children five years of age and under per household and village. A randomization ceremony for the intervention took place to randomly assign the villages to receive IRS or maintain their current status. Participants in both IRS and non-IRS areas were randomly chosen and consented to participate in cohorts to be followed prospectively. The total population disaggregated in under five years of age and above five in each village in the district will be used as a denominator for the passive case detection component of the study. Each house was geopositioned during the census visit as part of the household enumeration for spraying. This information can assist in defining the cluster size, core and buffer areas. Each household will receive a unique permanent ID. This is an interventional study with IRS serving as the research intervention.

To determine the incidence by active case detection, a cohort of children five years of age and under will be followed monthly from the core zone of each cluster. During each visit the care taker will answer a short questionnaire regarding health, net usage and health-related expenditure. The temperature of each recruited child will be recorded and an RDT performed. If the child has a positive RDT, irrespective of accompanying clinical symptoms he/she will receive treatment according to the national guidelines.

At health facility level, a separate facility-based team will ensure the collection of the household location (village) of each malaria case to determine the incidence in the different study clusters by passive case detection. Joint work with the community health workers (Agentes Polivantes Elementares [APEs]) will also strengthen quality of their data and they will be asked to include information on the location (village) of each malaria case they diagnose/treat.

Costing data will be prospectively collected using standardized data collection tools to determine the cost of interventions (IRS and LLIN distribution) and of care-seeking.

Cross-sectional studies will be carried out at the peak of transmission season in 2017, 2018, and 2019. There is a potential for the monthly visits for active case detection to have an influence on household behavior and expenditure. Additional data on house expenditure will be collected during the cross-sectionals to assess societal costs of malaria care that is independent from study visits.

Entomological data including mosquito densities, sporozoite rates, resistance status and indoor/outdoor biting ratios will be sampled from IRS and non-IRS villages throughout the study following standard PMI procedures.

ELIGIBILITY:
Inclusion Criteria:

* all consenting adults, assenting minors (12-18) and caregivers of children under 12

Exclusion Criteria:

* all infants 0-6 months of age

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3915 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Cost per case averted in children five years of age and under at health facility level by adding Actellic-IRS | 24 months
  Incidence at health facility level by passive case detection (with enhanced surveillance and quality control) along with implementation costing data using an ingredients approach

SECONDARY OUTCOMES:
Entomological Indicators | 24 months
  Entomological measurements including descriptions of vector densities, estimates of human biting rates, sporozoite rates, measures of indoor and outdoor feeding behaviors, insecticide resistance patterns and estimates of entomological inoculation rates (EIR)
Parasite prevalence | 12 months
  Changes in community-based parasitaemia measured through cross-sectional surveys
Health Behavior | 24 months
  Changes in malaria avoidance and health seeking behavior through cohort surveys and cross-sectional surveys
Cost per malaria case averted in children five years of age and under at the community | 24months
  Derived from incidence in children five years of age and under at the community levels by active case detection along with implementation costing data using an ingredients approach

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Saute, Md, MSc, PhD, Principal Investigator — Centro de Investigacoes de Manhica; Molly Robertson, MA, MPH, Principal Investigator — PATH; Carlos Chaccour, MD, MSc, PhD, Principal Investigator — Barcelona Institute for Global Health; Rose Zulliger, PhD, Principal Investigator — US Presidents Malaria Initiative, Centers for Disease Control and Prevention; Abuchama Saifodine, PhD, Principal Investigator — US Presidents Malaria Initiative, USAID
Locations (2):
- Molly Robertson, Washington D.C., District of Columbia, United States
- Centro de Investigacoes de Manhica, Manhiça, Maputo Province, Mozambique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alonso S, Chaccour CJ, Wagman J, Candrinho B, Muthoni R, Saifodine A, Saute F, Robertson M, Zulliger R. Cost and cost-effectiveness of indoor residual spraying with pirimiphos-methyl in a high malaria transmission district of Mozambique with high access to standard insecticide-treated nets. Malar J. 2021 Mar 10;20(1):143. doi: 10.1186/s12936-021-03687-1. PMID 33691706
- [Derived] Chaccour C, Zulliger R, Wagman J, Casellas A, Nacima A, Elobolobo E, Savaio B, Saifodine A, Fornadel C, Richardson J, Candrinho B, Robertson M, Saute F. Incremental impact on malaria incidence following indoor residual spraying in a highly endemic area with high standard ITN access in Mozambique: results from a cluster-randomized study. Malar J. 2021 Feb 10;20(1):84. doi: 10.1186/s12936-021-03611-7. PMID 33568137
- [Derived] Wagman JM, Varela K, Zulliger R, Saifodine A, Muthoni R, Magesa S, Chaccour C, Gogue C, Tynuv K, Seyoum A, Dengela D, Saute F, Richardson JH, Fornadel C, Linton YM, Slutsker L, Candrinho B, Robertson M. Reduced exposure to malaria vectors following indoor residual spraying of pirimiphos-methyl in a high-burden district of rural Mozambique with high ownership of long-lasting insecticidal nets: entomological surveillance results from a cluster-randomized trial. Malar J. 2021 Jan 21;20(1):54. doi: 10.1186/s12936-021-03583-8. PMID 33478533
- [Derived] Chaccour CJ, Alonso S, Zulliger R, Wagman J, Saifodine A, Candrinho B, Macete E, Brew J, Fornadel C, Kassim H, Loch L, Sacoor C, Varela K, Carty CL, Robertson M, Saute F. Combination of indoor residual spraying with long-lasting insecticide-treated nets for malaria control in Zambezia, Mozambique: a cluster randomised trial and cost-effectiveness study protocol. BMJ Glob Health. 2018 Jan 30;3(1):e000610. doi: 10.1136/bmjgh-2017-000610. eCollection 2018. PMID 29564161